CLINICAL TRIAL: NCT02028052
Title: Procedural Outcomes in Endobronchial Ultrasound - Transbronchial Needle Aspiration (EBUS-TBNA) With and Without Rapid On-Site Evaluation (ROSE) by Cytopathologist
Brief Title: Procedural Outcomes in Endobronchial Ultrasound - Transbronchial Needle Aspiration (EBUS-TBNA) With and Without Rapid On-Site Evaluation (ROSE)
Acronym: ROSE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: similar study data published
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00036432
Record Dates: First submitted 2013-12-20; First posted 2014-01-06 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2015-01

CONDITIONS: ENDOBRONCHIAL ULTRASOUND - TRANSBRONCHIAL NEEDLE ASPIRATION; Benign and Malignant Mediastinal and Hilar Lymph Nodes Known or Suspected Malignancy
Keywords: enlarged mediastinal nodes; enlarged hilar lymph nodes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ROSE (Other): In the case of ROSE, sampling frequency will occur similarly, but no additional samples will be taken in the case of provision of a preliminary diagnosis.
  Interventions: Procedure: ROSE; Device: 22 gauge Vizishot needles
- NO ROSE (Other): In the case of no ROSE, sampling frequency will be predetermined at 4 needle aspirations per site
  Interventions: Procedure: ROSE; Device: 22 gauge Vizishot needles

INTERVENTIONS:
Procedure: ROSE — The procedure will proceed with conventional EBUS-TBNA sampling of the target lesion with 22 gauge Vizishot needles. Each subject will be randomized to either ROSE by cytopathologist or no ROSE.
Device: 22 gauge Vizishot needles

SUMMARY:
The objective of this study is comparing the attributable procedural time of Endobronchial Ultrasound - Transbronchial Needle Aspiration (EBUS-TBNA) when sampling mediastinal and hilar lymph nodes with or without Rapid On-Site Evaluation (ROSE). The primary outcome will be the time elapsed from EBUS bronchoscope insertion to bronchoscope withdrawal. Secondary outcomes will include total number of sampled lymph nodes, average number of needle aspirations per lymph node sampled, overall diagnostic yield, and procedural time of the cytopathologist.

ELIGIBILITY:
Inclusion Criteria:

1. Subject provides informed consent
2. Subject is >18 years of age
3. Subject is scheduled to undergo flexible bronchoscopy with EBUS-TBNA of suspected enlarged mediastinal or hilar lymph nodes as part of their standard medical care
4. A negative pregnancy test in women of child-bearing potential
5. Subject is mentally capable of following study directions

Exclusion Criteria:

1. Study subject has any disease or condition that interferes with safe completion of initial or follow-up assessments
2. Concurrent participation in another study involving investigational drugs or investigational medical devices
3. Inability to read and understand the necessary study documents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Time lapse | during procedure, approximately 45 minutes
  The primary endpoint is the time elapsed from EBUS bronchoscope insertion to bronchoscope withdrawal.

SECONDARY OUTCOMES:
Total number of sampled lymph nodes | approximately 45 minutes
  Samples taken during procedure
Average number of needle aspirations per lymph node sampled | approximately 45 minutes
  Determined by tumor
Overall diagnostic yield | approximately 45 minutes
Procedural time of the cytopathologist | approximately 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Momen Wahidi, MD, MBA, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Yasufuku K, Chiyo M, Sekine Y, Chhajed PN, Shibuya K, Iizasa T, Fujisawa T. Real-time endobronchial ultrasound-guided transbronchial needle aspiration of mediastinal and hilar lymph nodes. Chest. 2004 Jul;126(1):122-8. doi: 10.1378/chest.126.1.122. PMID 15249452
- [Background] Mejia CP. [Surgery and orthodontics in the treatment of unerupted maxillary cuspids]. Rev Fed Odontol Colomb. 1976 Jan-Jun;24(116-117):47-52. No abstract available. Spanish. PMID 1076725
- [Background] Griffin AC, Schwartz LE, Baloch ZW. Utility of on-site evaluation of endobronchial ultrasound-guided transbronchial needle aspiration specimens. Cytojournal. 2011;8:20. doi: 10.4103/1742-6413.90081. Epub 2011 Nov 21. PMID 22145008
- [Background] Layfield LJ, Bentz JS, Gopez EV. Immediate on-site interpretation of fine-needle aspiration smears: a cost and compensation analysis. Cancer. 2001 Oct 25;93(5):319-22. doi: 10.1002/cncr.9046. PMID 11668466